CLINICAL TRIAL: NCT06219278
Title: A Retrospective Review Evaluating the Matrix Pro Applicator for Treatment of Wrinkles
Status: Completed | Type: Observational
Sponsor: Candela Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MXP23001
Record Dates: First submitted 2023-12-21; First posted 2024-01-23 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Wrinkle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Matrix Pro Applicator: Source study subjects received up to three (3) full-face treatments for wrinkles with Matrix Pro Applicator (27W)
  Interventions: Device: Profound Matrix

INTERVENTIONS:
Device: Profound Matrix — The source study consisted of up to three treatment visits with treatment intervals 6 weeks ± 2 weeks

SUMMARY:
This is a retrospective chart review of data from the multi-site prospective clinical trial, "Functional Usability and Feasibility Testing of the Profound Matrix™ System (FUFT2002)" to evaluate the safety and efficacy of the Profound Matrix System Matrix Pro applicator for the treatment of wrinkles.

DETAILED DESCRIPTION:
This was a retrospective medical record review of subject data from the source study FUFT2002 to evaluate the safety, efficacy, tolerability, and usability of the Profound MatrixTM System with the Matrix Pro Applicator for the treatment of wrinkles.

ELIGIBILITY:
Inclusion Criteria:

1. Met eligibility criteria under source study FUFT2002 and enrolled into FUFT2002 study (NCT # pending).
2. Received full face treatment with 27W Matrix Pro applicator only.
3. Have baseline and follow-up assessments obtained.
4. Have photography obtained with the VISIA standardized camera system (Appendix III).

Exclusion Criteria:

1. Sun exposure during the course of the study.
2. Aesthetic procedures and/or treatments during the course of the study.
3. Any violation of study treatment instructions.
4. Upon inspection, any differences in baseline and follow up photos that would not make evaluation of photos viable (e.g. chin placement, facial expression).
5. Any protocol deviation or change in study visit activities that would jeopardize reliability or validity of the retrospective review

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data was extracted from the records of 32 subjects previously enrolled in the source study who satisfied current study eligibility criteria, were aged 25-70 years, with Fitzpatrick Skin Types II-IV and had received full face treatments with the 27W Matrix Pro Applicator
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2023-10-29 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konika Patel Schallen, MD, Principal Investigator — Candela Medical
Locations (2):
- Candela Institue for Excellence, Marlborough, Massachusetts, United States
- Syneron Medical, Yokneam Illit, Israel

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Matrix Pro Applicator
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Matrix Pro Applicator
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.53 (10.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 29
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 19
  Israel | 13

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Facial Wrinkles
Description: Improvement in the appearance of wrinkles was assessed by three (3) blinded evaluators comparing photographs taken at Baseline/Pre-treatment and at the 3-month follow-up (post final treatment). Success for an individual subject (an individual responder) was determined if at least two out of three evaluators correctly identified the post-treatment photograph by selecting the correct corresponding photograph side (left or right).
Time Frame: Approximately 6 months following baseline assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Matrix Pro Applicator
Number analyzed (Participants) | 32
Participants | 24

2. Secondary Outcome: Subject Global Aesthetic Improvement Scale (GAIS)
Description: Assessment of Subject Assessment of Improvement via GAIS ratings at the study endpoint (3MFU) using a 5-point scale (-1= worse to 3= very much improved)
Time Frame: Approximately 6 months following baseline assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Matrix Pro Applicator
Number analyzed (Participants) | 32
Participants
  Very Much Improved | 4
  Much Improved | 13
  Improved | 13
  No Change | 2
  Worse | 0

3. Secondary Outcome: Subject Global Aesthetic Improvement Scale (SGAIS)
Description: Assessment of Subject Assessment of Improvement via GAIS ratings at a study timepoint using a 5-point scale (-1= worse to 3= very much improved)
Time Frame: Approximately 4 months following baseline assessment
Population: data was not collected and analyzed for this outcome
Arm/Group | Matrix Pro Applicator
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for approximately 3 years from initiation of source study on October 27, 2020, until completion of this retrospective analysis on July 1, 2024.
Arm/Group | Matrix Pro Applicator
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 5/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Matrix Pro Applicator (N=32)
Swelling (Immune system disorders) | 1 (1) — Experienced swelling as suspected allergic reaction to an unknown allergen.
Irregular Cardiac Rhythm (Cardiac disorders) | 1 (1) — Experienced ?irregular cardiac rhythms via smartwatch and was evaluated by a cardiologist. Determined not related to study procedures
Itchy bumps on skin (Skin and subcutaneous tissue disorders) | 1 (1)
Herpetic Outbreak (Immune system disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) — Closed, dry wound on the submentum and erythema in the right nasolabial folds following Tx. 1 complicated by subject picking at skin.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/78/NCT06219278/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-13): https://cdn.clinicaltrials.gov/large-docs/78/NCT06219278/SAP_001.pdf